CLINICAL TRIAL: NCT05760677
Title: Study on the Efficacy and Safety of Chiglitazar Sodium in the Treatment of Polycystic Ovary Syndrome With Type 2 Diabetes
Brief Title: Study on the Efficacy and Safety of Chiglitazar Sodium in PCOS With T2DM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chiglitazar sodium
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-02

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; T2D
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pioglitazone group (Active Comparator): All participants were treated with lifestyle intervention+ metformin(0.5g bid po)+ orlistat (0.12g bid po) (obese patients)+ pioglitazone (15mg qd po)
  Interventions: Drug: pioglitazone group: lifestyle intervention+ metformin+ orlistat (obese patients)+ pioglitazone; Drug: the Chiglitazar group: lifestyle intervention+ metformin+ orlistat (obese patients)+ Chiglitazar
- Chiglitazar group (Experimental): All participants were treated with lifestyle intervention+ metformin(0.5g bid po)+ orlistat (0.12g bid po) (obese patients)+ Chiglitazar (32mg QD)
  Interventions: Drug: pioglitazone group: lifestyle intervention+ metformin+ orlistat (obese patients)+ pioglitazone; Drug: the Chiglitazar group: lifestyle intervention+ metformin+ orlistat (obese patients)+ Chiglitazar

INTERVENTIONS:
Drug: pioglitazone group: lifestyle intervention+ metformin+ orlistat (obese patients)+ pioglitazone — the pioglitazone group： classic treatment: lifestyle intervention+ metformin+ orlistat (obese patients)+ pioglitazone
Drug: the Chiglitazar group: lifestyle intervention+ metformin+ orlistat (obese patients)+ Chiglitazar — the Chiglitazar group: lifestyle intervention+ metformin+ orlistat (obese patients)+ Chiglitazar (32mg QD)

SUMMARY:
Purpose and significance: To explore the clinical efficacy and safety of Chiglitazar sodium in polycystic ovary syndrome with type 2 diabetes

Methods: From October 2022 to September 2024, a total of 142 PCOS with T2DM patients admitted to Department of Endocrinology and Metabolism at the Affiliated Hospital of Nantong University were recruited. Participants are randomized in a ratio of 1:1 into two treatment groups of 71 participants: ① control group；②experimental group. After randomization, the control group was treated with lifestyle intervention+ metformin+ orlistat (obese patients)+ pioglitazone, and the patients in the experimental group were treated with lifestyle intervention+ metformin+ orlistat (obese patients)+ Chiglitazar (32mg QD) until the end of follow-up. The treatment and follow-up period totaled 3 months. Observe the body weight, menstrual cycle and blood glucose control and other related indicators.

Type of study: randomized controlled, prospective, intervention study.

DETAILED DESCRIPTION:
From October 2022 to September 2024, a total of 142 PCOS with T2DM patients admitted to Department of Endocrinology and Metabolism at the Affiliated Hospital of Nantong University were recruited. Participants are randomized in a ratio of 1:1 into two treatment groups of 71 participants: ① control group；②experimental group. After randomization, the control group was treated with lifestyle intervention+ metformin+ orlistat (obese patients)+ pioglitazone, and the patients in the experimental group were treated with lifestyle intervention+ metformin+ orlistat (obese patients)+ Chiglitazar (32mg QD) until the end of follow-up. The treatment and follow-up period totaled 3 months. Observe the body weight, menstrual cycle and blood glucose control and other related indicators.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Type 2 diabetes mellitus Clinical diagnosis of Polycystic ovarian syndrome Must be able to swallow tablets

Exclusion Criteria:

Mental diseases, autoimmune diseases, hematological diseases, malignant tumors, other ovarian diseases (such as ovarian cysts), sexually transmitted diseases Infertility caused by gynecological diseases such as uterine cat's eye disease and other reasons Abnormal function of important organs Congenital adrenocorticosis, hypothyroidism, Cushing's syndrome and other endocrine diseases Patients who have recently prepared or become pregnant

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of plasma glucose | 12 weeks
  Assessment the change level of plasma glucose. The unit is mmol/L.
The recovery of menstrual cycle | 12 weeks
  Assessment the recovery of menstrual cycle. The unit is day.

SECONDARY OUTCOMES:
The changes in body weight | 12 weeks
  Assessment the changes of body weight. The unit is kilogram.

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yunjuan, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided